CLINICAL TRIAL: NCT03345355
Title: MRI of Sacroiliac Joints: Evaluation of Accuracy of Dixon Sequences in the Diagnosis of Axial Spondyloarthritis
Acronym: SPADIX
Status: Terminated | Type: Observational
Why Stopped: Departure of the project leader
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/AL-01
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with axial spondyloarthritis
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — Coronal oblique T1, Coronal oblique and axial STIR, Coronal oblique T1 Dixon, Coronal oblique and Axial T2 Dixon and T1 Dixon post Gadolinium

SUMMARY:
The investigators hypothesize that the T1 Dixon post-Gadolinium and T2 Dixon sequences will show good diagnostic performances for active sacroiliitis compared to the reference test (Short tau inversion recovery) and clinical-biological criteria, which will allow a better diagnosis of active sacroiliitis

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient has a clinically diagnosed axial spondyloarthritis (axSpA) (ASAS or AMOR classification)
* Patient has an active axSpA (BASDAI>4)

Exclusion Criteria:

* The subject is participating in another study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding
* The patient has a contra-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically-confirmed axial spondyloarthritis treated in the radiology services of the CHUs of Montpellier and Nimes
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of T1 Dixon post-Gadolinium and T2 Dixon for active sacroiliitis, according to subchondral edema status | Time 0
  compared to ASAS criteria incorporating Short tau inversion recovery and clinic-biological elements

SECONDARY OUTCOMES:
Diagnosis of enthesitis from T1 Gadolinium Dixon sequence vs ASAS criteria | Time 0
  Yes/no
Diagnosis of synovitis from T2 Dixon and T1 Gadolinium Dixon sequences vs ASAS criteria | Time 0
  Yes/no
Diagnosis of chronic sacroiliite (erosion or chondral scler osis, or fatty spinal replacement) by T1 Dixon pre-Gadolinium | Time 0
  Yes/No
Diagnosis of chronic sacroiliite (erosion or chondral sclerosis, or fatty spinal replacement) by conventional sequences | Time 0
  Yes/no

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Lapeyronie, Montpellier
  - CHU Nimes, Nîmes